CLINICAL TRIAL: NCT04972604
Title: CureDuchenne Link®: A Resource to Support Research Studies in Duchenne and Becker Muscular Dystrophy (DMD/BMD)
Brief Title: CureDuchenne Link®: A Resource for Research
Acronym: CDLink
Status: Recruiting | Type: Observational
Sponsor: CureDuchenne (Other)
Responsible Party: Sponsor
Other Study IDs: CD-2021-01
Record Dates: First submitted 2021-06-21; First posted 2021-07-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Carrier; DMD; BMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, Urine, Saliva, Muscle and Skin will be collected. Sample collection will be optional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Duchenne and Becker muscular dystrophy: Individuals with Duchenne muscular dystrophy and Becker muscular dystrophy
- Carriers: Carriers of Duchenne muscular dystrophy and Becker muscular dystrophy

SUMMARY:
CureDuchenne link is a data hub comprised of integrated biospecimens, clinical data, and self- and/or caregiver-reported information from participants. Anyone over 4 weeks old who has been diagnosed with DMD or BMD or who is a carrier of DMD or BMD can join. Parents or legal guardians can sign up their child(ren).

DETAILED DESCRIPTION:
Individuals can participate through the CureDuchenne Link™ application (accessible via mobile device or web interface) and receive communications about research opportunities and community programs. Participation may be done using virtual methods, at a project site, and/or at community events nationwide.

All collected information will be stored in a secure, HIPAA-compliant data warehouse for approved researchers to use for studies relevant to DMD, BMD and other neuromuscular disorders. Combining health and outcomes data with biospecimens provides an impactful solution and novel resource for researchers, allowing for effective translational research.

ELIGIBILITY:
Inclusion Criteria:

1. Any of the following are true:

   1. Currently has a confirmed diagnosis of DMD/BMD based on genetic testing, muscle biopsy, or clinical diagnosis.
   2. Currently has a confirmed diagnosis of carrier status for DMD/BMD based on genetic testing.
2. Parent/guardian (for minor participants) or participant gives informed consent and/or assent as required by local regulations.
3. Is age 4 weeks or older at the time of consent.

Exclusion Criteria:

1. Is a foster child or ward of the state.
2. Is a prisoner.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with or carriers of Duchenne muscular dystrophy (DMD) and Becker muscular dystrophy (BMD).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2031-07-09 (Estimated); Study Completion 2031-07-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | Upon study entry
  There is no intervention in this project. Participants will provide documentation to support their diagnosis of Duchenne muscular dystrophy, Becker muscular dystrophy, or a carrier of these mutations
Genetic Mutation | Upon study entry or when genetic testing results are available
  Participants will be asked to provide genetic testing reports confirming their diagnosis, where available, which will be reviewed by a central genetic counselor.

SECONDARY OUTCOMES:
Functional Status | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Self reported data (questionnaire on ambulation and mobility) will be captured
North Star Ambulation Assessment (NSAA) Score | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Clinically reported NSAA scores will be captured
6 Minute Walk Test (6MWT) Score | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Clinically reported 6MWT scores will be captured
Corticosteroid Status | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Self reported and clinically reported corticosteroid status (past and present) will be captured
Cardiac Status | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Self reported and clinically reported cardiac status (past and present) will be captured
Respiratory Status | Upon study entry and every 6-12 months thereafter for up to ten (10) years
  Self reported and clinically reported respiratory status (past and present) will be captured

CONTACTS AND LOCATIONS:
Overall Officials: Debra Miller, Principal Investigator — CureDuchenne
Locations (10):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - CureDuchenne, Newport Beach, California
  - Children's Hospital of Orange County, Orange, California
  - Rare Disease Research, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Kansas University Clinical Research Center, Fairway, Kansas
  - Corewell Health, Grand Rapids, Michigan
  - Rare Disease Research Center, Hillsborough, North Carolina
  - Penn State Health, Hershey, Pennsylvania
  - Neurology Rare Disease Center, Denton, Texas

IPD SHARING:
Plan to Share IPD: Yes
After a thorough application process, data will be shared to qualified researchers.
  Approved researchers will complete all required CDA/data transfer agreements with CureDuchenne. Once complete, they will be given access to a limited dataset with direct identifiers removed.

REFERENCES:
- See also: CureDuchenne Link Information Page — https://www.cureduchenne.org/cureduchenne-link/